CLINICAL TRIAL: NCT04262089
Title: Neo-adjuvant Pembrolizumab in dMMR/ POLE-EDM Uterine Cancer Patients: a Feasibility Study
Acronym: PAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hans W. Nijman, MD PHD, Principal Investigator, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAM-UMCG-001
Record Dates: First submitted 2020-01-28; First posted 2020-02-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Uterine Cancer
Keywords: Uterine cancer; dMMR; POLE-EDM; neo-adjuvant; pembrolizumab
MeSH Terms: conditions — Uterine Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: A window-of-opportunity study of ICB in primary dMMR UC (n=10) and primary POLE-EDM UC (n=10) patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- primary dMMR uterine cancer patients (Experimental): primary dMMR uterine cancer patients
  Interventions: Drug: Pembrolizumab (Keytruda)
- primary POLE-EDM uterine cancer patients (Experimental): primary POLE-EDM uterine cancer patients
  Interventions: Drug: Pembrolizumab (Keytruda)

INTERVENTIONS:
Drug: Pembrolizumab (Keytruda) — Pembrolizumab (Keytruda), 200mg IV Q3W for a total of 2 administrations per patient, integrated into standard-of-care protocol prior to surgery. Based on the well-established time lines, the interval between diagnosis and standard of care hysterectomy is sufficient to treat patients with two cycles of pembrolizumab without interfering with standard of care.

SUMMARY:
In this feasibility study the investigators intend to treat patients with high mutational uterine cancer with two cycles immune checkpoint inhibition before standard-of-care hysterectomy.

DETAILED DESCRIPTION:
Objective:

The investigators aim to establish proof-of-concept for use of immune checkpoint blockade (ICB) as novel neo-adjuvant therapy in (deficient mismatch repair) dMMR and (Polymerase ε mutation)POLE-EDM uterine cancer (UC). When ICB proves to be feasible as defined in the primary endpoint, a follow-up with a larger multicenter studies to determine clinical efficacy, such as postponing standard-of-care surgery or randomized studies to standard-of-care.

Study design:

The investigators planned a window-of-opportunity study of ICB in primary dMMR UC (n=10) and primary POLE-EDM UC (n=10) patients. ICB (pembrolizumab; anti-PD1) will be administered in two cycles of 3 weeks between diagnosis and standard-of-care hysterectomy.

Tumor responses to pembrolizumab will be assessed 3 weeks after the second cycle of pembrolizumab by a pathologist (primary endpoint) and MRI (secondary endpoint).After treatment with immun checkpoint blockade a hysterectomy will take place (standard-of care). Peripheral blood and tumor samples will be used to evaluate immune responses.

Study population:

Primary dMMR/ POLE-EDM UC patients of any stage and/or grade who are intended to be treated with a hysterectomy recruited from the North-Netherlands oncological region.

Intervention: Pembrolizumab, 200mg IV Q3W for a total of 2 administrations per patient, integrated into standard-of-care protocol prior to surgery. Based on the well-established time lines, the interval between diagnosis and standard of care hysterectomy is sufficient to treat patients with two cycles of pembrolizumab without interfering with standard of care.

Main study endpoints:

The primary endpoint is the response rate of the tumor assessed by pathology in uterine cancer patients treated with neo-adjuvant pembrolizumab. The secondary endpoint is the objective response rate of the tumor by MRI using RECIST. Exploratory objectives are immunogenicity, safety and the value of a pipelle biopsy as a predictor for response.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed primary diagnosis of dMMR/POLE-EDM uterine cancer who are intended to be treated with hysterectomy will be enrolled in this study.
* Have measurable disease based on RECIST 1.1 on MRI.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, is not a woman of childbearing potential (WOCBP) or agrees to follow the contraceptive guidance in section 5.2 during the treatment period and at least until standard-of-care hysterectomy.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation.

Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.

* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to characterize pathologic responses (necrosis/viable tumor cells) in uterine cancer patients treated with neo-adjuvant pembrolizumab | Tumor tissue is collected during standard of care hysterectomy (up to 6-10 weeks after baseline)
  Hematoxylin and eosin staining on endometrium tissue collected during standard-of-care hysterectomy will be assessed by an experienced pathologist for evidence of necrosis and/or viable tumor cells
The primary objective is to characterize pathologic responses (Degree of immune infiltration) in uterine cancer patients treated with neo-adjuvant pembrolizumab | Tumor tissue is collected during standard of care hysterectomy (week 6-10 after baseline)
  Hematoxylin and eosin staining on endometrium tissue collected during standard-of-care hysterectomy will be assessed by an experienced pathologist for degree of immune infiltration.
The primary objective is to characterize pathologic responses (Degrees of inflammation, fibrosis, and mucin) in uterine cancer patients treated with neo-adjuvant pembrolizumab | Tumor tissue is collected during standard of care hysterectomy (week 6-10 after baseline)
  Hematoxylin and eosin staining on endometrium tissue collected during standard-of-care hysterectomy will be assessed by an experienced pathologist for degrees of inflammation, fibrosis, and mucin, consistent with an ongoing immune response.

SECONDARY OUTCOMES:
Radiologic response | MRI is scheduled before start study drug (week 1) and after final study drug ( 6-10 weeks after baseline)
  To assess the objective response rate of the tumor by MRI using RECIST1.1 in uterine cancer patients treated with 2 cycles neo-adjuvant pembrolizumab

OTHER OUTCOMES:
Systemic immune response using an IFN-y-ELISPOT to screen for the presence of antigen-specific T-cell responses to mutation associated neo antigens | At 6 timepoints through the study up to 32 weeks.
  Collection of PBMC (60mL blood by vena puncture) before, during and after treatment to assess antigen specific T cell responses to mutation-associated neo-antigens
Safety (adverse events) | Through study completion, an average of 32 weeks.
  Adverse events will be documented according CTCAE.
Feasibility (surgical delays due to study treatment) | Up to planned hysterectomy (6-10 weeks after baseline)
  The number of treatment-related surgical postponements will be counted to assess feasibility.
Predictive value of pipelle biopsy | An additional pipelle biopsy is obtained before start of the hysterectomy (6-10 weeks after baseline).
  In order to assess the correlation of pathological response seen in the biopsy and the surgical specimen. A pipelle biopsy will be obtained during surgery and assess as the tumor specimen from hysterectomy in the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Hans W Nijman, Prof. Dr., Principal Investigator — University Medical Center Groningen, UMCG; An KL Reyners, Prof. Dr., Principal Investigator — University Medical Center Groningen, UMCG
Locations (1):
- Universitair Medisch Centrum Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eerkens AL, Brummel K, Vledder A, Paijens ST, Requesens M, Loiero D, van Rooij N, Plat A, Haan FJ, Klok P, Yigit R, Roelofsen T, de Lange NM, Klomp R, Church D, Ter Elst A, Wardenaar R, Spierings D, Foijer F, Koelzer VH, Bosse T, Bart J, Jalving M, Reyners AKL, de Bruyn M, Nijman HW. Neoadjuvant immune checkpoint blockade in women with mismatch repair deficient endometrial cancer: a phase I study. Nat Commun. 2024 Sep 3;15(1):7695. doi: 10.1038/s41467-024-52098-8. PMID 39227583